CLINICAL TRIAL: NCT04413344
Title: Double-Blind Comparative Trial and Open-Label Extension Trial to Investigate the Safety and Efficacy of TW-012R in Alzheimer's Disease With Presenilin 1 (PSEN1) Mutations
Brief Title: Repurposing Bromocriptine for Abeta Metabolism in Alzheimer's Disease
Acronym: REBRAnD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kyoto University (Other)
Collaborators: Mie University (Other); Osaka University (Other); Tokushima University (Unknown); Tokyo Metropolitan Institute for Geriatrics and Gerontology (Unknown); Asakayama Hospital (Unknown); Kawasaki Medical School Hospital (Unknown); Nagoya City University Hospital (Unknown); Time Therapeutics, Inc. (Unknown); Towa Pharmaceutical Co.,Ltd. (Unknown)
Responsible Party: Principal Investigator, Haruhisa Inoue, Professor, Kyoto University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IACT19029
Record Dates: First submitted 2020-05-28; First posted 2020-06-02 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Familial Alzheimer Disease (FAD); PSEN1 Mutation
MeSH Terms: conditions — Alzheimer Disease | interventions — Bromocriptine

STUDY DESIGN:
Intervention Model Description: [Double-blind phase] Multicenter, randomized, placebo-controlled, double-blind, parallel-group comparison clinical trial [Extension phase] Multicenter, open-label, extension trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Active Comparator): Bromocriptine mesilate, 2.5 to 22.5 mg per day, divided three times a day, for 50 weeks.
  Interventions: Drug: Bromocriptine Mesilate
- Placebo (Placebo Comparator): Placebo, divided three times a day, for 50 weeks.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Bromocriptine Mesilate — Each tablet contains 2.87 mg of bromocriptine mesilate (JP) (2.5 mg of bromocriptine)
  Other Names: TW-012R
  Arms: Active
Drug: Placebos — Identical tablets which contain no active ingredient
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn about safety and efficacy of bromocriptine in familial Alzheimer's disease with presenilin 1 mutations.

The main questions it aims to answer are: •safety of bromocriptine •efficacy of bromocriptine

Participants will answer questions, have blood exams, lumbar punctures and MRI/PET scans. Researchers will compare a participants group taking bromocriptine with a participants group taking placebo to see if there is any changes in cognitive function, and behavioral and psychiatric symptoms with dementia.

DETAILED DESCRIPTION:
To investigate the safety and efficacy of an orally administered dose of TW-012R in patients with Alzheimer's disease bearing PSEN1 (presenilin 1) mutations (PSEN1-AD), using a placebo group as a control. In addition, long-term safety will be examined in an open-label extension trial.

ELIGIBILITY:
Inclusion Criteria:

* Alzheimer's disease patients with PSEN1 mutations
* Patients diagnosed with "probable AD" according to the diagnostic guideline of NIA-AA or "probable Alzheimer-type dementia" according to the diagnostic criteria for Alzheimer's disease specified in DSM-5
* An MMSE-J score of <= 25
* Patients whose cognitive function and everyday function are obviously impaired based on their medical record or information provided by a person who knows the patient well
* Patients for whom intellectual disability and mental disorders other than dementia can be ruled out based on their academic background, work history, and life history.
* Patients with a reliable and close relationship with a partner/caregiver
* Age>=20 years at the time of giving informed consent
* Written informed consent has been obtained from the patient or his/her legally acceptable representative to participate in this trial

Exclusion Criteria:

* Difficulty with the oral intake of tablets
* Patients receiving anti-dementia drugs who have changed the dosing regimen during the 2 months prior to giving informed consent
* Patients with dementia due to pathology other than Alzheimer's disease (e.g., vascular dementia, frontotemporal dementia, Lewy body dementia, progressive supranuclear palsy, corticobasal degeneration, Huntington's disease, and prion disease)
* Presence of clinically relevant or unstable mental disorders. Patients with major depression in remission can be enrolled.
* Imminent risk of self-harm or harm to others
* Body mass index (BMI) of <= 17 or >= 35
* Patients with a history of alcohol dependence, drug dependence, or drug abuse within the 5 years before providing informed consent
* HBs antigen positive
* Anti-HIV antibody positive
* Anti-HTLV-1 antibody positive
* Patients with an active infection, such as hepatitis C and syphilis (STS/TPHA)
* Patients with the following liver function values on the test before enrollment
* AST(GOT) > 4.0 x Upper limit of the institutional reference range or
* ALT (GPT) > 4.0 x Upper limit of the institutional reference range
* Patients who have uncontrolled, clinically significant medical conditions (e.g., diabetes melitus, hypertension, thyroid/endocrine disease, congestive cardiac failure, angina pectoris, cardiac/gastrointestinal disease, dialysis, and abnormal renal function with an estimated CLcr < 30 mL/min)within 3 months prior to giving informed consent in addition to the underlying disease to be investigated in the trial and for whom the investigator or sub-investigator considers that there is a significant medical risk in the patient's participation in the trial
* Patients with long QT syndrome or tendency toward prolonged QTc interval (male: >=470 msec, female: >= 480 msec), or patients with a history/complication of torsades de pointes
* Patients with a history of malignancies within 5 years prior to providing informed consent. However, patients with the following diseases can be enrolled if they are treated appropriately:
* Skin cancer (basal cell, squamous cell)
* Cervical carcinoma in situ
* Localized prostate cancer
* Malignancies that have not recurred for at least 3 years since surgery and the patient's physician has determined that the risk of recurrence is low
* Patients with clinically significant vitamin B1/B12 deficiency or folic acid deficiency within 6 months prior to giving informed consent
* Patients who have participated in other clinical research/trials involving interventions within the 3 months prior to providing informed consent
* Patients who have previously received bromocriptine or TW-012R
* Patients with a history of hypersensitivity to bromocriptine or ergot alkaloids
* Patients with current or a history of thickened heart valve cusps, restricted heart valve motion, and the associated heart valve lesions, such as stenosis, confirmed by echocardiography
* Pregnant females, lactating females, females who may be pregnant, and females who wish to become pregnant
* Other patients who are considered inappropriate to participate in this trial at the discretion of the investigator or sub-investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
Safety (Incidence and severity of adverse events and adverse reactions) | Until Week 50 (end of trial)
  to assess safety
Severe impairment battery-Japanese version (SIB-J) | Until Week 20 and 36
  to assess cognitive function
Neuropsychiatric Inventory (NPI) | Until Week 20 and 36
  to assess behavioral and psychiatric symptoms of dementia

SECONDARY OUTCOMES:
Mental Function Impairment Scale (MENFIS) | Until Week 20 and 36
  to assess cognitive function
Mini-Mental State Examination-Japanese (MMSE-J) | Until Week 20 and 36
  to assess cognitive function
Disability Assessment for Dementia (DAD) | Until Week 20 and 36
  to assess activities of daily living
Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III | Until Week 20 and 36
  to assess motor symptoms and signs
Apathy Scale | Until Week 20 and 36
  to assess apathy
Plasma Aβ protein concentration | Until Week 20 and 36
  to assess Aβ protein metabolism
Plasma NfL protein concentration | Until Week 20 and 36
  to assess neurodegeneration
Plasma Total Tau, Plasma p-Tau concentration | Until Week 20 and 36
  to assess tau protein metabolism
Cerebrospinal fluid (CSF) Aβ concentration | Until Week 36
  to assess Aβ protein metabolism
CSF Total Tau, CSF p-Tau concentration | Until Week 36
  to assess tau protein metabolism
Blood bromocriptine concentration | Until Week 20 and 36
  to assess safety

OTHER OUTCOMES:
Wearable physical activity meter | Until Week 20 and 36
  to assess activities of daily living
Finger tapping sensor readout | Until Week 20 and 36
  to assess finger tapping
Brain amyloid PET image | Until Week 36
  to assess Aβ protein metabolism
Brain tau PET image | Until Week 36
  to assess tau protein metabolism
Upper motor neuron burden score | Until Week 20 and 36
  to assess spasticity
Plasma Aβ-related peptides concentration | Until Week 20 and 36
  to assess Aβ protein metabolism

CONTACTS AND LOCATIONS:
Overall Officials: Haruhisa Inoue, MD, PhD, Principal Investigator — Kyoto University; Hidekazu Tomimoto, MD, PhD, Study Director — Mie University Hospital; Haruhiko Banno, MD, PhD, Study Director — Kyoto University Hospital
Locations (8):
- Japan (8):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Kyoto University Hospital, Kyoto, Kyoto
  - Mie University Hospital, Tsu, Mie-ken
  - Kawasaki Medical School Hospital, Kurashiki, Okayama-ken
  - Asakayama Hospital, Sakai, Osaka
  - Osaka University, Suita, Osaka
  - Tokushima University Hospital, Tokushima, Tokushima
  - Tokyo Metropolitan Institute for Geriatrics and Gerontology, Tokyo, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Individual data from all the participants are illustrated in the figures and in appendix of journal article. Any data shown will be available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: After publication
Access Criteria: Reasonable request

REFERENCES:
- [Derived] Kondo T, Banno H, Okunomiya T, Amino Y, Endo K, Nakakura A, Uozumi R, Kinoshita A, Tada H, Morita S, Ishikawa H, Shindo A, Yasuda K, Taruno Y, Maki T, Suehiro T, Mori K, Ikeda M, Fujita K, Izumi Y, Kanemaru K, Ishii K, Shigenobu K, Kutoku Y, Sunada Y, Kawakatsu S, Shiota S, Watanabe T, Uchikawa O, Takahashi R, Tomimoto H, Inoue H. Repurposing bromocriptine for Abeta metabolism in Alzheimer's disease (REBRAnD) study: randomised placebo-controlled double-blind comparative trial and open-label extension trial to investigate the safety and efficacy of bromocriptine in Alzheimer's disease with presenilin 1 (PSEN1) mutations. BMJ Open. 2021 Jun 30;11(6):e051343. doi: 10.1136/bmjopen-2021-051343. PMID 34193504